CLINICAL TRIAL: NCT05964907
Title: Optimizing Phototesting and Investigating Photobiology of Visible Light
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Indermeet Kohli, Associate Scientist, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14869
Record Dates: First submitted 2023-04-19; First posted 2023-07-28 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- VL+UVA1 (Other): Participants will be treated with VL + UVA1 light source
  Interventions: Device: Light Source B: Visible Light solar simulator (VL + UVA1); Device: Light Source A: Visible Light solar simulator closer match to sunlight (VL +UVA1)

INTERVENTIONS:
Device: Light Source B: Visible Light solar simulator (VL + UVA1) — Patients will be radiated with light source B (Visible light solar simulator)
Device: Light Source A: Visible Light solar simulator closer match to sunlight (VL +UVA1) — Patients will be radiated with light source A (Visible light solar simulator closer match to sunlight)

SUMMARY:
Specific Aim 1: To determine the impact of spectral composition of the VL+UVA1 source on the associated biologic effects.

Specific Aim 2: To investigate differential responses of subjects with different skin phototypes to VL+UVA1, including immediate and delayed erythema and pigmentation, and photodamage.

DETAILED DESCRIPTION:
The design of the study consists of a total of 4 visits within a two week period. The first visit consists of VL+UVA1 irradiation with different light source on the opposite site of patients' back. A combination of non-invasive measurements (e.g., photography, redness and color changes of the skin using colorimetry and diffuse reflectance spectrometry) will be conducted throughout the 4 visits. Biopsies will be taken at various time points.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals age 18 and older
* Fitzpatrick skin phototype (SPT) I-VI, 7 with SPT I-III and 7 with SPT IV-VI, with normal healthy skin
* Able to understand the requirements of the study and its associated risks
* Able to complete and sign a consent form
* Willing and able to refrain from any medications or herbal supplements during the duration of the study, unless permitted by the investigator
* Agrees to refrain from using any new topical skin care products, laundry detergents, or fragrances while participating in the study
* Has not had excessive sun exposure for 7 days prior to enrollment in the study

Exclusion Criteria:

* Recent history of vitiligo, melasma, and other disorders of pigmentation with the exception of post-inflammatory hyperpigmentation
* History of relevant skin conditions such as atopic dermatitis, eczema, or sunburn on any part of the body
* History of photodermatoses or photosensitivity disorders
* History of melanoma or non-melanoma skin cancers
* Use of tanning parlors or exposure of the irradiated sites to sun light during the duration of the study
* Use of topical or systemic treatment that is likely to interfere with assessment, study results, or pose safety concerns
* Subjects with a tendency to bleed excessively
* Known allergies to anesthetics (lidocaine) or anaphylaxis treatment (epinephrine)
* History of hypertrophic scarring or keloid formation
* Use of any photosensitizing medication within the visible light range or additional medication at the discretion of the investigator [examples include - but not limited to - thiazide diuretics, regular use of NSAIDs, hydroxychloroquine, or voriconazole
* A woman who is lactating, pregnant, or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Erythema assessment for all 14 participants. | Visit 1 (Day 0)
  Measured clinically with Investigator Global Assessment (IGA) scale IGA Description of Erythema (Redness) 0 Clear of erythema
  1. Almost clear of erythema
  2. Mild, but noticeable erythema
  3. Moderate erythema (pink), no sharp borders
  4. Severe erythema (dark pink), sharp borders
  5. Very severe erythema (very dark pink to almost red)
Erythema assessment for all participants | Visit 2 (Day 1)
  Measured clinically with Investigator Global Assessment (IGA) scale IGA Description of Erythema (Redness) 0 Clear of erythema
  1. Almost clear of erythema
  2. Mild, but noticeable erythema
  3. Moderate erythema (pink), no sharp borders
  4. Severe erythema (dark pink), sharp borders
  5. Very severe erythema (very dark pink to almost red)
Erythema assessment | Visit 3 (Day 7)
  Measured clinically with Investigator Global Assessment (IGA) scale IGA Description of Erythema (Redness) 0 Clear of erythema
  1. Almost clear of erythema
  2. Mild, but noticeable erythema
  3. Moderate erythema (pink), no sharp borders
  4. Severe erythema (dark pink), sharp borders
  5. Very severe erythema (very dark pink to almost red)
Erythema assessment for 14 participants | Visit 4 (Day 14)
  Measured clinically with Investigator Global Assessment (IGA) scale IGA Description of Erythema (Redness) 0 Clear of erythema
  1. Almost clear of erythema
  2. Mild, but noticeable erythema
  3. Moderate erythema (pink), no sharp borders
  4. Severe erythema (dark pink), sharp borders
  5. Very severe erythema (very dark pink to almost red)
Erythema assessment for all 14 participants | Visit 1 (Day 0)
  Both colorimetry and DRS non-invasively provide quantitative objective information regarding changes in skin color by quantifying skin hyperpigmentation and erythema as L* and a* by colorimeter, and as melanin, oxy-hemoglobin concentration by DRS respectively. ITA can be derived from L* and b* by using ITA = [arctan (L* - 50)/b*] X 180/Π)].
  Colorimetry: Decrease in L* and ITA indicates greater pigmentation. Increase in a* indicates increase in Erythema. All these parameters are relative with arbitrary units DRS: Increase in Melanin content will indicate increase in pigmentation and increase in oxy-hemoglobin will indicate increase in erythema. All these parameters are relative with arbitrary units
Erythema assessment for all 14 participants | Visit 2 (Day 1)
  Both colorimetry and DRS non-invasively provide quantitative objective information regarding changes in skin color by quantifying skin hyperpigmentation and erythema as L* and a* by colorimeter, and as melanin, oxy-hemoglobin concentration by DRS respectively. ITA can be derived from L* and b* by using ITA = [arctan (L* - 50)/b*] X 180/Π)].
  Colorimetry: Decrease in L* and ITA indicates greater pigmentation. Increase in a* indicates increase in Erythema. All these parameters are relative with arbitrary units DRS: Increase in Melanin content will indicate increase in pigmentation and increase in oxy-hemoglobin will indicate increase in erythema. All these parameters are relative with arbitrary units
Erythema assessment for all 14 participants | Visit 3 (Day 7)
  Both colorimetry and DRS non-invasively provide quantitative objective information regarding changes in skin color by quantifying skin hyperpigmentation and erythema as L* and a* by colorimeter, and as melanin, oxy-hemoglobin concentration by DRS respectively. ITA can be derived from L* and b* by using ITA = [arctan (L* - 50)/b*] X 180/Π)].
  Colorimetry: Decrease in L* and ITA indicates greater pigmentation. Increase in a* indicates increase in Erythema. All these parameters are relative with arbitrary units DRS: Increase in Melanin content will indicate increase in pigmentation and increase in oxy-hemoglobin will indicate increase in erythema. All these parameters are relative with arbitrary units
Erythema assessment for all 14 participants | Visit 4 (Day 14)
  Both colorimetry and DRS non-invasively provide quantitative objective information regarding changes in skin color by quantifying skin hyperpigmentation and erythema as L* and a* by colorimeter, and as melanin, oxy-hemoglobin concentration by DRS respectively. ITA can be derived from L* and b* by using ITA = [arctan (L* - 50)/b*] X 180/Π)].
  Colorimetry: Decrease in L* and ITA indicates greater pigmentation. Increase in a* indicates increase in Erythema. All these parameters are relative with arbitrary units DRS: Increase in Melanin content will indicate increase in pigmentation and increase in oxy-hemoglobin will indicate increase in erythema. All these parameters are relative with arbitrary units
Pigmentation assessment for all 14 participants. | Visit 1 (day 0)
  Measured clinically with Investigator Global Assessment (IGA) scale IGA Description of Pigmentation (Tanning) 0 Clear of hyperpigmentation
  1. Almost clear of hyperpigmentation
  2. Mild, but noticeable hyperpigmentation
  3. Moderate hyperpigmentation (medium brown)
  4. Severe hyperpigmentation (dark brown)
  5. Very severe hyperpigmentation (very dark brown to almost black)
Pigmentation assessment for all 14 | Visit 2 (Day 1)
  Measured clinically with Investigator Global Assessment (IGA) scale IGA Description of Pigmentation (Tanning) 0 Clear of hyperpigmentation
  1. Almost clear of hyperpigmentation
  2. Mild, but noticeable hyperpigmentation
  3. Moderate hyperpigmentation (medium brown)
  4. Severe hyperpigmentation (dark brown)
  5. Very severe hyperpigmentation (very dark brown to almost black)
Pigmentation assessment for 14 participants | Visit 3 (Day 7)
  Measured clinically with Investigator Global Assessment (IGA) scale IGA Description of Pigmentation (Tanning) 0 Clear of hyperpigmentation
  1. Almost clear of hyperpigmentation
  2. Mild, but noticeable hyperpigmentation
  3. Moderate hyperpigmentation (medium brown)
  4. Severe hyperpigmentation (dark brown)
  5. Very severe hyperpigmentation (very dark brown to almost black)
Pigmentation assessment for all 14 | Visit 4 (Day 14)
  Measured clinically with Investigator Global Assessment (IGA) scale IGA Description of Pigmentation (Tanning) 0 Clear of hyperpigmentation
  1. Almost clear of hyperpigmentation
  2. Mild, but noticeable hyperpigmentation
  3. Moderate hyperpigmentation (medium brown)
  4. Severe hyperpigmentation (dark brown)
  5. Very severe hyperpigmentation (very dark brown to almost black)
Pigmentation assessment for all 14 participants.. | Visit 1 (day 0)
  Both colorimetry and DRS non-invasively provide quantitative objective information regarding changes in skin color by quantifying skin hyperpigmentation and erythema as L* and a* by colorimeter, and as melanin, oxy-hemoglobin concentration by DRS respectively. ITA can be derived from L* and b* by using ITA = [arctan (L* - 50)/b*] X 180/Π)].
  Colorimetry: Decrease in L* and ITA indicates greater pigmentation. Increase in a* indicates increase in Erythema. All these parameters are relative with arbitrary units DRS: Increase in Melanin content will indicate increase in pigmentation and increase in oxy-hemoglobin will indicate increase in erythema. All these parameters are relative with arbitrary units
Pigmentation assessment for all 14 participants | Visit 2 (Day 1)
  Both colorimetry and DRS non-invasively provide quantitative objective information regarding changes in skin color by quantifying skin hyperpigmentation and erythema as L* and a* by colorimeter, and as melanin, oxy-hemoglobin concentration by DRS respectively. ITA can be derived from L* and b* by using ITA = [arctan (L* - 50)/b*] X 180/Π)].
  Colorimetry: Decrease in L* and ITA indicates greater pigmentation. Increase in a* indicates increase in Erythema. All these parameters are relative with arbitrary units DRS: Increase in Melanin content will indicate increase in pigmentation and increase in oxy-hemoglobin will indicate increase in erythema. All these parameters are relative with arbitrary units
Pigmentation assessment for all 14 participants | Visit 3 (Day 7)
  Both colorimetry and DRS non-invasively provide quantitative objective information regarding changes in skin color by quantifying skin hyperpigmentation and erythema as L* and a* by colorimeter, and as melanin, oxy-hemoglobin concentration by DRS respectively. ITA can be derived from L* and b* by using ITA = [arctan (L* - 50)/b*] X 180/Π)].
  Colorimetry: Decrease in L* and ITA indicates greater pigmentation. Increase in a* indicates increase in Erythema. All these parameters are relative with arbitrary units DRS: Increase in Melanin content will indicate increase in pigmentation and increase in oxy-hemoglobin will indicate increase in erythema. All these parameters are relative with arbitrary units
Pigmentation assessment for all 14 participants | Visit 4 (Day 14)
  Both colorimetry and DRS non-invasively provide quantitative objective information regarding changes in skin color by quantifying skin hyperpigmentation and erythema as L* and a* by colorimeter, and as melanin, oxy-hemoglobin concentration by DRS respectively. ITA can be derived from L* and b* by using ITA = [arctan (L* - 50)/b*] X 180/Π)].
  Colorimetry: Decrease in L* and ITA indicates greater pigmentation. Increase in a* indicates increase in Erythema. All these parameters are relative with arbitrary units DRS: Increase in Melanin content will indicate increase in pigmentation and increase in oxy-hemoglobin will indicate increase in erythema. All these parameters are relative with arbitrary units

SECONDARY OUTCOMES:
Immunohistochemical changes in pigmentation, inflammation, and profileration, for all 14 participants | Visit 1 (Day 0)
  Histology assess parameter including pigmentation, inflammation and proliferation.
Immunohistochemical changes in pigmentation, inflammation, and profileration, for all 14 participants | Visit 2 (Day 1)
  Histology assess parameter including pigmentation, inflammation and proliferation.
Immunohistochemical changes in pigmentation, inflammation, and profileration, for all 14 participants | Visit 3 (Day 7)
  Histology assess parameter including pigmentation, inflammation and proliferation.
RNA sequencing for 8 participants | Visit 2 (Day 1)
  Molecular changes- sample collection for RNA sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Medical Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No